CLINICAL TRIAL: NCT04715360
Title: Management of Cytokine Storms in Severe COVID-19 Patients With Autologous Activated Platelet-rich Plasma Therapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hayandra Peduli Foundation (Other)
Collaborators: Koja Regional Public Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-12-1526
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Covid19; Sars-CoV-2 Infection; ARDS, Human; Severe covid19
Keywords: aaPRP; severe COVID-19; platelet-rich plasma; SARS-CoV-2; autologous
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome | interventions — favipiravir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Only received standard medication (avigan) for severe COVID-19 management
  Interventions: Drug: Avigan
- PRP Group (Experimental): received standard medication (avigan) for severe COVID-19 management and autologous activated platelet-rich plasma transfusion
  Interventions: Combination Product: autologous activated platelet-rich plasma; Drug: Avigan

INTERVENTIONS:
Combination Product: autologous activated platelet-rich plasma — Patient received standard medication for COVID-19 management and autologous activated platelet-rich plasma on day 1, 3 and 5 while patient in ICU. On day 0, 4 and 6, hematology analysis, multicytokines measurement and thorax X-ray were done to each patient
  Arms: PRP Group
Drug: Avigan — Patient received avigan 2x1,600 mg for a day, followed by 2x600 mg for five consecutive days.

SUMMARY:
The positive cases of coronavirus disease-2019 (COVID-19) in Indonesia has been increasing rapidly since the first case found in March 2020 to date. Coronavirus 2 (SARS-CoV-2) virus disrupts human normal immune system resulting in uncontrolled inflammatory response. Based on our research and experience in doing cell therapy for 9 years, activated platelet-rich plasma (PRP) produces anti-inflammatory effects in inflammatory condition that is beneficial for tissue regeneration. In this study, we aimed to evaluate the potential of autologous activated platelet-rich plasma (aaPRP) and the outcomes for treating severe Coronavirus Disease-2019 (COVID-19) patients in Intensive Care Unit (ICU).

DETAILED DESCRIPTION:
PRP decreases IL-1β, IL-6, IL-8, and TNFα inflammatory genes expression while also reduces IL-1β and TNFα inflammatory cytokines production. PRP has also been showed to contain interleukin 1 receptor antagonist (IL-1RA), an anti-inflammatory cytokines that suppress IL-6 secretion.

ELIGIBILITY:
Inclusion Criteria:

* severe covid-19 patient in ICU

Exclusion Criteria:

* CKD on hemodialysis, HIV positive, hepatitis, pregnant, destroyed lung, cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-29 (Actual); Primary Completion 2021-11-29 (Estimated); Study Completion 2021-12-27 (Estimated)

PRIMARY OUTCOMES:
Effect of aaPRP on pro-inflammatory cytokines plasma level (IL-6, IL-1B, TNFa, IFN gamma, MCP-1) before and after intervention compared to control. | 6 days
  Patients with positive COVID19 who will improve after receiving aaPRP compared to control.
to evaluate the change of Effect of aaPRP on anti-inflammatory cytokines plasma level (IL-1RA, IL-4, IL-10) before and after intervention compared to control. | 6 days
  Patients with positive COVID19 who will improve after receiving aaPRP compared to control.
Effect of aaPRP on overall adverse event related to the treatment. | 6 days
  Patients with positive COVID19 who will improve after receiving aaPRP compared to control.
Effect of aaPRP on CRP level before and after intervention compared to control. | 6 days
  Patients with positive COVID19 who will improve after receiving aaPRP compared to control.

SECONDARY OUTCOMES:
Effect of aaPRP on Thorax X-ray image pre and post intervention between control and aaPRP-treated group | 6 days
  Patients with positive COVID19 who will improve after receiving aaPRP compared to control.
Effect of aaPRP on duration of hospitality of patient compared to control | 6 days
  Patients with positive COVID19 who will improve after receiving aaPRP compared to control.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Martin Christoffel, MD, Principal Investigator — Koja Regional Public Hospital
Locations (1):
- Koja Regional Public Hospital, Jakarta, DKI Jakarta, Indonesia